CLINICAL TRIAL: NCT05229666
Title: Stress Phenotypes and Preterm Birth: Immune and Energetic Cellular Dysregulation and the Preventive Effect of Social Support
Brief Title: Stress Phenotypes and Preterm Birth
Acronym: PTB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Catherine Monk, Diana Vagelos Professor of Women's Mental Health (in Obstetrics and Gynecology and Psychiatry), Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAU9052; R01MD016278 (NIH); 8144 (Other: New York State Psychiatric Institute Institutional Review Board)
Record Dates: First submitted 2022-01-19; First posted 2022-02-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Preterm Birth; Inflammation; Stress; Mental Health Issue
MeSH Terms: conditions — Premature Birth; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Challenge (Other)
  Interventions: Other: Cognitive Challenge

INTERVENTIONS:
Other: Cognitive Challenge — Cognitive challenge delivered via computer.

SUMMARY:
Pregnancy ends in preterm birth (PTB) for approximately 1 in 10 women, though more often for Non-Hispanic Black women, 14.12% PTB rate, compared to 9.09% for Non-Hispanic White women. Psychosocial stress and childhood trauma each are associated with risk for PTB and PTB has an intergenerational impact: mothers born preterm are more likely to give birth pretern, especially amongst Black women. In this project, we will study mitochondria, which contain their own genome, the mitochondria DNA, and are inherited from the mother, as they represent a potential intersection point between psychosocial experiences and their biological embedding in underlying disease outcomes such as PTB

DETAILED DESCRIPTION:
At odds with common assumptions - and hope, pregnancy ends in preterm birth (PTB) for approximately 1 in 10 women. Yearly PTB affects 15 million infants worldwide and 386,580 in the United States. PTB is the leading cause of global, and U.S., neonatal mortality and morbidity and is associated with future risk for poor physical (higher blood pressure, chronic kidney disease, wheeze/asthma) and mental (ADHD, IQ decrements) health. Maternal health is not spared: women who deliver preterm are at an increased risk for depression, hypertension, cardiovascular and renal disease later in life. In the U.S., the racial and ethnic disparities in PTB rates are dramatic and independent of socio-economic status (SES): overall, 14.12% for Non-Hispanic Black compared to 9.09% for Non-Hispanic White women.

Psychosocial stress and childhood trauma each are associated with risk for PTB. PTB has an intergenerational impact: mothers born preterm are more likely to give birth pretern, especially amongst Black women. Biomarkers to predict PTB have proven unsuccessful, and do not account for this emerging recognition of intergenerational transmission of PTB risk specifically via maternal heritage. Mitochondria, which contain their own genome, the mitochondria DNA, are inherited from the mother and represent a potential intersection point between psychosocial experiences and their biological embedding, including via immune dysregulation, in underlying disease outcomes. We aim to apply a mitochondria psychobiology approach to delineate by which mechanisms life stress - including discrimination and childhood trauma - results in disproportionate risk of PTB in minority women, and evaluate mitochondria as potential biomarkers of this birth outcome.

In a sample of post-attrition n=175 pregnant women we will test the following three aims: Aim 1: To determine whether a data driven approach to multiple, 1st trimester psychosocial (self- report stress discrimination, 24-hour ambulatory mood, social support), lifecourse (hair cortisol, childhood trauma), and biological variables (acute laboratory physiological stress reactivity) generate unique stress profiles that partially explain the racial/ethnic differences in gestational age at birth. Aim 2: To identify molecular indices of mitochondrial and immune functioning in the mother (3x blood draw), placenta, and fetal cord blood that mediate the association between 1st trimester maternal stress phenotypes and risk for earlier gestational age at birth. Aim 3: To evaluate if reduction in stress levels and/or improvement in social support over the course of pregnancy is associated with molecular indices of mitochondrial and immune functioning and (exploratory) reduced risk of earlier birth relative to national and hospital norms.

This new conceptual framing of this adverse health outcome (1) incorporates evidence of the psychosocial factors contributing to risk, (2) aims to account for the racial/ethnic disparities, and (3) harnesses cutting-edge mitochondria knowledge and tools to better characterize PTB's pathophysiology and identify novel targets for its intervention and prevention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, singleton pregnancy, between the ages of 18-45

Exclusion Criteria:

* Currently smoking cigarettes, drinking alcohol, taking dugs, taking medications regularly (other than prenatal vitamins), multiple fetal pregnancy, inflammatory conditions including rheumatoid arthritis, lupus, and multiple sclerosis, and not planning to deliver at CUMC

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Higher percentage of Black and Hispanic women in high stress group | Between 36-38 weeks gestation
  The high stress group is calculated using various measures including multiple psychosocial, life course, biological variables, and acute stress reactivity to a cognitive challenge (Stroop test).

SECONDARY OUTCOMES:
Relatively earlier gestational age at birth in high stress group | At birth
  The high stress phenotype is calculated using various measures including, multiple psychosocial, life course, biological variables, and acute stress reactivity to a cognitive challenge (Stroop test).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No